CLINICAL TRIAL: NCT04947462
Title: Proprioceptive Sensorimotor Integration With Neural Interfaces for Hand Prostheses
Acronym: PSI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: A3699-R; RX003699-01 (Other Grant/Funding Number: VA RR&D); 1624763-1 (Other: IRBNET)
Record Dates: First submitted 2021-06-23; First posted 2021-07-01 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Upper Limb Amputees
Keywords: Proprioception; Prosthesis; Upper Extremity Limb Loss; Peripheral Nerve Stimulation; Embodiment; Sensorimotor; Neuroprostheses

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Chronically Implanted Neural and Muscular Interface (Experimental): 6 eligible participants will be chronically implanted with neural and muscular interfaces to characterize proprioceptive sensations using Functional Electrical Stimulation (FES).
  Interventions: Device: Chronically Implanted Neural and Muscular Interface

INTERVENTIONS:
Device: Chronically Implanted Neural and Muscular Interface — Participants will be chronically implanted with neural and muscular interfaces to characterize proprioceptive sensations using Functional Electrical Stimulation (FES).

SUMMARY:
The purpose of this study is to characterize proprioceptive sensations in the missing limb of upper limb amputees using nerve stimulation, and to develop advanced controllers for moving a prosthesis. Proprioceptive sensations are the sensations that tell individuals where their hand is in space, and if it is moving. The research team uses Functional Electrical Stimulation (FES), which involves applying small electric currents to the nerves. These signals are then transferred to the brain just like the information about the individual's intact hand used to be transferred to their brain. This study will test different placements for stimulation and determine which one(s) provide the individual with proprioceptive sensations. The investigators want to know what the participants feel and if the investigators can use proprioceptive sensation to give the participants information about limb movement and position.

DETAILED DESCRIPTION:
Hands are the primary means of interacting with the world, and Veterans who have lost a hand must cope with diminished functional and sensory capabilities. While myoelectric prostheses can restore the basic grasping function of the lost hand, many amputees abandon use of prostheses because current prosthetic options do not meet their needs. In addition, many amputees struggle with phantom pain and psychosocial deficits following limb loss that are not fully mitigated by current treatments.

In the normal sensorimotor system, proprioception, which is the sense of limb position and movement, is critical for informing motor plans and correcting errors in movement. In addition, proprioception plays a key role in body ownership, agency, and phantom pain. Despite its importance, proprioception is absent in current prosthetic options.

The goal of the proposed project is to make upper limb prosthetic devices more natural and useful for Veterans who have lost a hand by providing proprioceptive feedback about prosthesis postures and movements. The central hypothesis is that effectively closing the loop between a prosthesis user and their device requires that the sensory inputs and control outputs closely mimic the underlying sensorimotor neural processes of the body schema. The investigators will examine integration of artificial proprioception with prosthesis control in three trans-radial and three trans-humeral amputees using the investigators' implanted neural-interfacing system.

Aim 1. Characterize proprioceptive sensations elicited by peripheral nerve stimulation. The investigators will test time-varying Peripheral Nerve Stimulation (PNS) patterns and examine the impact on the kinematics of the evoked proprioceptive percept using position matching with the contralateral intact limb and multivariate regression analyses. The investigators will investigate paired agonist-antagonist stimulation strategies and compare the discriminability between agonist-only and paired agonist-antagonist strategies using psychometric tests.

Aim 2. Investigate the mechanisms of stimulation-evoked proprioception. The neurophysiological basis of proprioception from PNS is unknown. To investigate whether proprioceptive percepts originate from direct afferent activation or indirect recruitment via direct muscle activation, the investigators will perform a motor block of the residual forearm of trans-radial participants and examine changes to the proprioceptive percepts. In trans-humeral participants, Targeted Muscle Reinnervation will be performed at the time of system implant, and percepts will be compared before and after muscle ingrowth.

Aim 3. Determine the integration of proprioceptive stimulation with motor control during posture matching. To restore proprioception to Veterans during active prosthesis use, PNS-evoked percepts must be integrated with voluntary limb control. The investigators will determine the impact of proprioception on motor control through a virtual reality posture matching task and compare performance with velocity and position-based prosthetic hand controllers with and without proprioceptive PNS. Second, the investigators will determine the impact of voluntary control on the perception of PNS-evoked proprioception through a psychometric dissimilarity rating task. Third, the investigators will assess the impact of artificial proprioception on embodiment via surveys.

The project will be the first to investigate the sensorimotor integration of proprioception from PNS in a broad population of upper-limb amputees and with both position and velocity controllers. The study will provide important information about the kinematics of artificial proprioception and the role of direct muscle activation in forming proprioceptive percepts. The investigators expect that knowledge gained in this proposal will improve prosthesis utility and acceptance for Veterans with limb loss and will advance prosthetic hand technology and standard of care in the neurorehabilitation field.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral upper limb amputation above or below the elbow with fully healed and healthy surgical sites
* Viable peripheral nerve function in the residual nerves serving the limb
* Volitional activity of the residual muscles in the amputated limb or actuating movement of the limb
* Medically fit to undergo general anesthesia
* Fitted with a prosthesis by a certified prosthetic and orthotic specialist (CPO) and at least one month of experience using a prosthesis
* Willingness and availability to follow the study protocol
* Willingness to undergo psychological evaluation, if recommended by study surgeons or investigators, to determine that the participant is mentally competent and capable of completing the study-related activities

Exclusion Criteria:

* Bilateral upper limb amputation, unless the amputation on the contralateral side only involves missing digits but does not qualify as a partial hand amputation
* Inability to speak English
* Medically unfit to undergo surgery
* Pregnancy, or those who are of childbearing potential, unwilling to prevent pregnancy during the trial
* Uncontrolled diabetes (HgbA1c>8.0%)
* History of neuropathy and/or radiculopathy in the target limb
* Active infection or open sores on the residual limb
* History of frequent infection or sores with unknown cause
* Inability to provide informed consent or follow experimental protocols
* Severe pain that would prevent the participant from completing study-related activities
* Poor surgical candidate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Magnitude of change in perceived joint position | This metric will be measured approximately each month for two years.
  Magnitude of change in perceived joint position, as measured by joint angle transducers in the Cyberglove.

CONTACTS AND LOCATIONS:
Overall Officials: Emily L Graczyk, PhD, Principal Investigator — Louis Stokes VA Medical Center, Cleveland, OH
Locations (1):
- Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: E. Gardner, J. Martin, in Principles of neural science (2000; — https://www.semanticscholar.org/paper/Coding-of-Sensory-Information-Gardner-Martin/331c40a1ae5ca02446b4234653dcfd289c4e1b44?p2df